CLINICAL TRIAL: NCT00005401
Title: Validation and Exploration of Sleep and Mood Predictors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4318; R01HL055983 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-07

CONDITIONS: Sleep Apnea Syndromes; Depression; Lung Diseases; Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes; Depression; Lung Diseases

SUMMARY:
To determine whether objectively recorded sleep durations were mortality risk factors, whether sleep duration could be distinguished from depression as a risk factor in Women's Health Initiative (WHI) data, and whether sleep-associated risks were attributable to specific pathophysiologic processes such as sleep apnea, circadian rhythm phase advances, or deficiencies of melatonin, or deficiencies of reproductive steroids. The study was ancillary to the WHI.

DETAILED DESCRIPTION:
BACKGROUND:

Both reported short sleep and reported long sleep are major predictors of excess mortality risk, but the importance of reported sleep duration as a risk factor is not yet known. Sleep-related risks are of special interest to The Women's Health Initiative (WHI), because insomnia increases among women at menopause, and because WHI's hormone replacement therapy (HRT) and dietary modification (DM) may influence sleep. The WHI is an exciting opportunity to examine whether risks associated with reported sleep durations can be explained by a selection of intercurrent conditions, but the broad WHI design does not control for important potential confounders. Explicitly, the broad WHI design by itself cannot determine if behaviorally-modifiable objective sleep durations are the primary risk factor.

DESIGN NARRATIVE:

This ancillary project supplemented the WHI Observational Study (OS) by performing additional examinations on 600 San Diego OS women. These volunteers underwent home sleep recordings, hormone measurement, and detailed psychiatric interviews. To facilitate distinction of affective and sleep factors in WHI outcomes, the types and severity of depression in the OS subsample and the validity and reliability of sleep items in questionnaires given to WHI women were examined.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-08; Study Completion 1999-07

REFERENCES:
- [Background] Kripke DF, Elliot JA, Youngstedt SD, Smith JS. Melatonin: marvel or marker? Ann Med. 1998 Feb;30(1):81-7. doi: 10.3109/07853899808999388. PMID 9556093
- [Background] Kripke DF, Klauber MR, Wingard DL, Fell RL, Assmus JD, Garfinkel L. Mortality hazard associated with prescription hypnotics. Biol Psychiatry. 1998 May 1;43(9):687-93. doi: 10.1016/s0006-3223(97)00292-8. PMID 9583003
- [Background] Kripke DF. Light treatment for nonseasonal depression: speed, efficacy, and combined treatment. J Affect Disord. 1998 May;49(2):109-17. doi: 10.1016/s0165-0327(98)00005-6. PMID 9609674
- [Background] Jean-Louis G, Kripke DF, Assmus JD, Langer RD. Sleep-wake patterns among postmenopausal women: a 24-hour unattended polysomnographic study. J Gerontol A Biol Sci Med Sci. 2000 Mar;55(3):M120-3. doi: 10.1093/gerona/55.3.m120. PMID 10795722
- [Background] Jean-Louis G, Kripke DF, Ancoli-Israel S, Klauber MR, Sepulveda RS, Mowen MA, Assmus JD, Langer RD. Circadian sleep, illumination, and activity patterns in women: influences of aging and time reference. Physiol Behav. 2000 Jan;68(3):347-52. doi: 10.1016/s0031-9384(99)00186-9. PMID 10716544
- [Background] Jean-Louis G, von Gizycki H, Zizi F. Predictors of subjective sleepiness induced by melatonin administration. J Psychosom Res. 1999 Oct;47(4):355-8. doi: 10.1016/s0022-3999(98)00076-2. PMID 10616229
- [Background] Jean-Louis G, Mendlowicz MV, Von Gizycki H, Zizi F, Nunes J. Assessment of physical activity and sleep by actigraphy: examination of gender differences. J Womens Health Gend Based Med. 1999 Oct;8(8):1113-7. doi: 10.1089/jwh.1.1999.8.1113. PMID 10565670
- [Background] Lasko TA, Kripke DF, Elliot JA. Melatonin suppression by illumination of upper and lower visual fields. J Biol Rhythms. 1999 Apr;14(2):122-5. doi: 10.1177/074873099129000506. PMID 10194648
- [Background] Jean-Louis G, Zizi F, von Gizycki H, Hauri P. Actigraphic assessment of sleep in insomnia: application of the Actigraph Data Analysis Software (ADAS). Physiol Behav. 1999 Jan 1-15;65(4-5):659-63. doi: 10.1016/s0031-9384(98)00213-3. PMID 10073464